CLINICAL TRIAL: NCT03870594
Title: Intradialytic Hypotension in Diabetic Haemodialysis Patients and Its Association With Dialytic Age
Brief Title: IDH in Diabetic Haemodialysis Patients and Association With Dialytic Age
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mahmoud Mohamed Fawzy (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Mohamed Fawzy, resident doctor at health insurance hospital ,Assiut, Egypt, Assiut University
Organization: Assiut University (Other)
Other Study IDs: IDH in diabetic patients
Record Dates: First submitted 2019-03-05; First posted 2019-03-12 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Intra-dialytic Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- diabetic: patients suffer from diabetes mellitus
  Interventions: Diagnostic Test: glycated hemoglobin
- non diabetic: patients free from diabetes with normal blood glucose level
  Interventions: Diagnostic Test: glycated hemoglobin

INTERVENTIONS:
Diagnostic Test: glycated hemoglobin — hemoglobin A1c level in blood

SUMMARY:
Intradialytic hypotension (IDH ) is a serious and the most frequent complication of hemodialysis of the hemodialysis .Diabetes is associated with autonomic neuropathy which contribute to intradialytic hypotension

DETAILED DESCRIPTION:
Intradialytic hypotension (IDH ) is a serious and the most frequent complication of hemodialysis of the hemodialysis.Intradialytic hypotension is a decrease in systolic BP by ≥20 mm Hg or a decrease in mean arterial pressure of 10 mm Hg associated with symptoms like cramps, dizziness, headache ,nausea and vomiting according to The National Kidney Foundation.Intradialytic hypotension occurs during 20%-30% of hemodialysis sessions. It is associated with poor long-term outcomes. Patients with Intradialytic hypotension show increased morbidity and mortality.The etiology of Intradialytic hypotension is multifactorial and depends on patient-related factors, as well as on complications related to the dialysis procedure. The main causes Intradialytic hypotension have been reported to be acute hypovolemia during ultrafiltration and inadequate compensatory mechanisms such as left ventricular dysfunction, inappropriate plasma refilling ,Impaired vasoconstriction induced by dysregulation of autonomic nervous system.

Diabetes mellitus is the most common cause of chronic renal failure .Diabetic patients are more prone to cardiovascular diseases than non-diabetics .Although diabetes is in relation with hypertension ,It is associated with autonomic neuropathy which contribute to intradialytic hypotension . Recent researches suggested that older age and long dialytic age may incease risk of intradialytic hypotension.

ELIGIBILITY:
Inclusion Criteria:

All haemodialysed end stage kidney disease patients of the haemodialysis unit in Assiut health insurance hospital

Exclusion Criteria:

* 1-Advanced heart failure 2-Clinical instability requiring hospital admission. 3-History of alcohol or substance abuse 4-previous history of psychotic disorders

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: all haemodialysed end stage kidney disease patients of the haemodialysis unit in Assiut health insurance hospital
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-04 (Estimated); Primary Completion 2019-06 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
the correlation between diabetes and intradialytic hypotension | 4 weeks
  Blood samples will be obtained for glycated hemoglobin, fasting blood glucose.Then patients will be divided into two groups DM, non DM.
  Blood pressure will be measured with mercury sphygmomanometer before, after and every 60 min during the hemodialysis session (a total of 5 measurements), for 10 consecutive dialysis sessions.Intradialytic hypotension (IDH) will defined as a decrease in systolic BP by ≥20 mm Hg or a decrease in mean arterial pressure of 10 mm Hg associated with symptoms
the correlation between dialytic age and intradialytic hypotension | 4 weeks
  Prior to the dialysis session,full history taking including age,duration of haemodialysis Blood pressure (BP) will be measured with mercury sphygmomanometer before, after and every 60 min during the hemodialysis session (a total of 5 measurements), for 10 consecutive dialysis sessions.
  Intradialytic hypotension (IDH) will defined as a decrease in systolic BP by ≥20 mm Hg or a decrease in mean arterial pressure of 10 mm Hg associated with symptoms